CLINICAL TRIAL: NCT03604926
Title: Immunophenotyping of Metastases From Colorectal Cancer
Status: Completed | Type: Observational
Sponsor: Istituto Oncologico Veneto IRCCS (Other)
Collaborators: Azienda Ospedaliera di Padova (Other); Azienda ULSS 16 Padova (Other)
Responsible Party: Sponsor
Other Study IDs: Take five
Record Dates: First submitted 2018-02-28; First posted 2018-07-30 (Actual); Last update posted 2020-11-20 (Actual); Status verified 2020-11

CONDITIONS: Metastatic Colorectal Cancer
MeSH Terms: conditions — Colorectal Neoplasms

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- chemo-naive patients
- pre-treated patients with systemic chemotherapy +/- a targeted

SUMMARY:
Immune therapy represents a promising option for the treatment of an increasing number of malignancies. New immunotherapeutic strategies are currently under development and will be further studied starting from refractory settings of heavily pre-treated mCRC patients. On this basis, a specific immunological characterization of CRC metastasis will be relevant to direct future clinical and pharmacological research.

As surgery is a therapeutic option in the treatment of mCRC, a percentage of mCRC patients undergo to resection of metastasis before or after medical treatment. These tumour samples could be useful to define the immune signature of colorectal metastatic disease.

On the basis of the above reported considerations, an exploratory, prospective, observational study for the immunophenotypical characterization of colorectal cancer metastasis from pre-treated vs chemo-naive patients has been planned.

DETAILED DESCRIPTION:
* There is extensive evidence for molecular heterogeneity in CRC. Studies have revealed that intra-tumour heterogeneity can be highly variable within primary tumours or between primary and metastatic sites (1). Moreover, tumour heterogeneity can be linked to targeted therapies in terms of acquired resistance mutations (2). In the era of precision medicine, specific molecular characterization of primary tumour and metastasis taking into account the dynamism of the disease and the actual therapeutic target should be considered.
* Nowadays there is not enough information regarding the immunological characterization of CRC metastasis. Especially, few data are available about the effect of chemotherapy and targeted drugs on the interplay between tumour and the immune system of the host (3).
* Immune system takes part to different phases of tumour growth (4). It is a dynamic balance that can be differentially modulated by several agents, resulting in immunosuppression or immunostimulation. Becht et al. integrated the molecular classification of colorectal cancer with information about their immune microenvironment. They identified 2 "immune-high subgroups". The MSI-rich CMS1 group is characterized by an immune stimulating contexture while the mesenchymal CMS4 group has an immune suppressive microenvironment (5). No data regarding the evolution over time of these features are available so far.
* Immune therapy represents a promising option for the treatment of an increasing number of malignancies. New immunotherapeutic strategies are currently under development and will be further studied starting from refractory settings of heavily pre-treated mCRC patients. On this basis, a specific immunological characterization of CRC metastasis will be relevant to direct future clinical and pharmacological research.
* As surgery is a therapeutic option in the treatment of mCRC, a percentage of mCRC patients undergo to resection of metastasis before or after medical treatment. These tumour samples could be useful to define the immune signature of colorectal metastatic disease.

On the basis of the above reported considerations, an exploratory, prospective, observational study is planned for the immunophenotypical characterization of colorectal cancer metastasis from pre-treated vs chemo-naive patients.

ELIGIBILITY:
Inclusion Criteria:

* Histological diagnosis of colorectal cancer
* Metastatic disease
* Surgery for metastatic disease
* Availability of clinical data

Exclusion Criteria:

* Non-metastatic disease

Sex: All
Age Groups: Child, Adult, Older Adult
Study Population: Pre-treated or chemo-naive patients with resected CRC metastasis
Sampling Method: Probability Sample
Enrollment: 10 (Actual)
Dates: Start 2017-10-05 (Actual); Primary Completion 2019-09-15 (Actual); Study Completion 2019-09-15 (Actual)

PRIMARY OUTCOMES:
immunological features of metastasis | through study completion, an average of 1 year
  Tumor-infiltrating lymphocytes (TIL)

CONTACTS AND LOCATIONS:
Locations (1):
- Istituto Oncologico Veneto IRCCS, Padua, Italy